CLINICAL TRIAL: NCT05807373
Title: Differential Diagnosis Between Parkinson's Disease and Multiple System Atrophy Using Digital Speech Analysis - Part 2 - Voice4PD-MSA-II
Brief Title: Differential Diagnosis Between Parkinson's Disease and Multiple System Atrophy Using Digital Speech Analysis - Part 2
Acronym: Voice4PD-MSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2016/34
Record Dates: First submitted 2023-03-24; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease; Multiple System Atrophy
Keywords: Motor speech disorder; dysarthria; speech processing; Parkinson's disease; Multiple System Atrophy
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parkinson's disease (Experimental): Diagnosis of idiopathic Parkinson's disease (PD) according to MDS criteria (Postuma et al., 2015)
  Interventions: Procedure: voice recordings
- Multiple system atrophy parkinsonian subtype (MSA-P) (Experimental): Diagnosis of Multiple Atrophy System (MSA-P) Parkinsonian form possible or probable according to consensus criteria (Gilman et al., 2008)
  Interventions: Procedure: voice recordings
- Healthy volunteer (Experimental): Absence of neurologic and oto-rhino-laryngologic disease
  Interventions: Procedure: voice recordings

INTERVENTIONS:
Procedure: voice recordings — A digital processing of voice recordings (from 30 to 45 minutes) will be performed for each participant, using a high quality digital recorder: the DIANA (computerized device of acoustic analysis) and the EVA-2 workstations (assisted Evaluation system Voice)

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease. Multiple system atrophy (MSA) is a relentlessly progressing rare neurodegenerative disease of unknown etiology. The differential diagnosis between the MSA-Parkinsonism (MSA-P) subtype and PD can be very challenging in early disease stages, while early diagnostic certitude is important for the patient because of the diverging prognosis. At the time being, there exists no validated objective biomarker to guide the clinician. Dysarthria is a common early symptom in both diseases and of different origin. The ambition and the originality of this project are to develop a digital voice-based tool for objective discrimination between PD and MSA-P.

DETAILED DESCRIPTION:
The team will build a corpus of voice samples of patients with both diseases and healthy volunteers. This corpus will consist of sustained vowels, pseudo-words, repetition of syllables, utterances of a standard text and spontaneous speech. Voice recordings will be performed using a high quality digital recorder (H4n) and the EVA-2 workstations. EVA-2 is a state-of-the-art system dedicated to pathological voice recording and analysis, which also allows the measurement of aerodynamic features such as intra-oral and subglottal pressure.

An electroglottograph (EGG), a non-invasive device, will also be used in conjunction with the recordings to provide the ground truth of glottal opening and closure instants (OGI and GCI) during utterances. The use of an EGG can be very useful given that OGI and GCI provide valuable information about the voice short-time dynamics.

The team will also perform a laryngostroboscopic examination to highlight defects in vocal cord mobility, a defect in vocal cord mating in phonation, abnormal vocal cord movements or supraglottic structures.

The primary objective is to compare a global score assessing vocal performance between MSA-P, PD and healthy volunteers. Secondary objectives are 1) to compare an acoustic index, assessing the subsystems of speech production, between MSA-P, PD and healthy volunteers, 2) to compare an acoustic index, assessing types of dysarthria, between MSA-P and PD patients, and 3) to compare perceptual assessment, performed by a panel of experts, of voice alteration between MSA-P and PD patients.

The final goal of this study is to evaluate the validity of the vocal markers that were identified in the previous study (Voice4PD-MSA-I, exploratory cohort). The validation will only consider data collected in the present study in order to assess the performance of the classifiers developed in the exploratory cohort.

ELIGIBILITY:
* Inclusion criteria:

  * Age from 30 to 80 years old
  * Signed informed consent
  * Affiliated to social security
  * Patient with PD :

    * Diagnosis of idiopathic Parkinson's disease (PD) according to criteria (Postuma et al., 2015)
    * Patient PD : Hoehn&Yahr stage between 1 and 2
    * Patient with or without mild to moderate speech troubles: MDS-UPDRS III item 1 ≤ 2
  * Patients with MSA-P :

    * Diagnosis of Multiple Atrophy System (MSA) Parkinsonian form possible or probable according to current consensus criteria (Gilman et al., 2008)
    * Patient MSA-P: score of part IV of the UMSARS ≤ 3 points
    * Patient with or without mild to moderate speech troubles: UMSARS II item 2 ≤ 2
  * Controls :

    * Absence of neurologic and oto-rhino-laryngologic disease
* Exclusion criteria :

  * Deafs and/or mutes
  * Patient with speech disorders which are not related to MSA or PD
  * Person under safeguard justice, guardianship

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-01-02 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of global vocal performance score based on six acoustic components | Day 1
  1. Differences between groups (PD, MSA-P, and controls) in global vocal performance score based on six acoustic components (1. Incoordination of articulatory movements: TDV (pseudowords), 2. Difficulty initiating movements: VOT (diadochokinesis), DPI (reading text and monologue), 3. Hyperkinetic movements: stdF0, stdPSD, DVA (held vowel /a/), 4. Reduced range of motion: stdF0 (read text and monologue), 5. Slowness of movement: NSR (read text), DDKR (diadochokinesis), VD (diadochokinesis), and 6. Irregularity of movements: DDKI (diadochokinesis)).

SECONDARY OUTCOMES:
measurements of a composite acoustic index assessing speech production subsystems | Day 1
  Differences between groups (PD, MSA-P, and controls) in a composite acoustic index, assessing speech production subsystems. The acoustic index will be calculated by linear combinations, described in [Daoudi et al., 2022], of features evaluating the performance of subsystems of speech production: breathing, phonation, articulation, prosody and timing.
measurements of a composite acoustic index assessing hypokinetic, ataxic and spastic dysarthria | Day 1
  Differences between groups (PD and MSA-P) in a composite acoustic index assessing hypokinetic, ataxic and spastic dysarthria. The acoustic index will be calculated by linear combinations, described in [Daoudi et al., 2022], of features assessing hypokinetic, ataxic and spastic dysarthria.
measurements of a vocal impairment score based on perceptual assessment by an expert jury (Range 1-10) | Day 1
  Differences between groups (PD and MSA-P) in a vocal impairment score based on perceptual assessment by an expert jury (Range 1-10). The score between 1 (for inaudible voice) and 10 (for normal voice) is calculated by averaging the sub-scores (between 1 and 10) evaluating intelligibility, articulation, prosody and resonance.

CONTACTS AND LOCATIONS:
Overall Officials: Wassilios MEISSNER, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Khalid DAOUDI, PhD, Study Chair — nstitut National de Recherche en Informatique et en Automatique
Locations (2):
- France (2):
  - CHU de Bordeaux - Institut des maladies neurodégénératives de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No